CLINICAL TRIAL: NCT00003138
Title: Phase III Evaluation of EPO With or Without G-CSF Versus Supportive Therapy Alone in the Treatment of Myelodysplastic Syndromes
Brief Title: Erythropoietin (EPO)+/- Filgrastim (G-CSF) vs. Supportive Therapy Alone for Patients With Myelodysplastic Syndromes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000065907; E1996 (Other: Eastern Cooperative Oncology Group (ECOG)); U10CA021115 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2013-12-06 (Estimated); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Anemia; Myelodysplastic Syndromes
Keywords: anemia; refractory anemia; myelodysplastic syndromes; erythropoietin; filgrastim
MeSH Terms: conditions — Anemia; Myelodysplastic Syndromes; Anemia, Refractory | interventions — Erythropoietin; Filgrastim; Granulocyte Colony-Stimulating Factor; Blood Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Supportive Care (Active Comparator): Patients received red cell and platelet transfusions for symptoms or to maintain hematocrit at or above 25% by volume. Patients who required transfusion support for symptomatic anemia prior to entering the study and who developed an increase in their transfusion requirement of >= 50% shall cross over to the Erythropoietin treatment arm, after at least four months on the supportive therapy arm.
  Interventions: Procedure: Transfusion
- Erythropoietin (Experimental): Erythropoietin was administered at 150 units/kg subcutaneously every day. If patients stopped responding, they were subsequently treated with Erythropoietin (150 units/kg) and filgrastim and then Erythropoietin (300 units/kg) and filgrastim.
  Interventions: Biological: Erythropoietin; Biological: Filgrastim

INTERVENTIONS:
Biological: Erythropoietin — Administered at 150 units/kg subcutaneously every day. Rotating sites should be used. The dose should be rounded off to the nearest 1000 U. The dose should be adjusted based on hematocrit.
  Other Names: r-HuEPO; EPO
  Arms: Erythropoietin
Biological: Filgrastim — G-CSF should start at a dose of 1 mcg/kg per day or 2.5 mcg/kg three times a week subcutaneously. Rotating sites should be used The dose should be rounded off to the nearest 10 mcg.
  Other Names: G-CSF; Neupogen; Recombinant-methionyl human granulocyte colony-stimulating factor; Granulocyte colony-stimulating factor; r-methHuG-CSF
  Arms: Erythropoietin
Procedure: Transfusion — Red cell and platelet transfusions
  Arms: Supportive Care

SUMMARY:
RATIONALE: Erythropoietin and colony-stimulating factors such as filgrastim stimulate the production of blood cells. It is not yet known whether erythropoietin with or without filgrastim is more effective than standard blood transfusions in reducing the need for transfusions in patients who have anemia associated with myelodysplastic syndrome.

PURPOSE: Randomized phase III trial to compare the effectiveness of erythropoietin with or without filgrastim with that of standard blood transfusions in reducing the need for transfusions in patients who have anemia associated with myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the benefit of erythropoietin vs standard transfusion support in reducing transfusion requirements in patients with myelodysplastic syndromes.
* Compare the clinical response, disease progression, and survival in patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.
* Evaluate whether adding filgrastim (G-CSF) or increasing the erythropoietin dose will reduce the transfusion requirement in patients who do not respond to erythropoietin alone.
* To compare the benefit of erythropoietin versus supportive care alone on quality of life (QOL) in persons with myelodysplastic syndromes.

OUTLINE: This is a randomized, controlled, multicenter, cross-over study. Patients are stratified according to morphologic subtype (refractory anemia [RA] vs RA with ringed sideroblasts vs RA with excess blasts), transfusion requirement (yes vs no), prior erythropoietin treatment (yes vs no), and erythropoietin level (at least 200 mU/mL vs less than 200 mU/mL). Patients are randomized to one of two treatment arms.

* Arm I (standard transfusion support): Patients receive red cell and platelet transfusions for symptoms or to maintain hematocrit level of 25% or above. Patients undergo bone marrow aspirate and biopsy at 4 months and then every year until development of acute leukemia or completion of study. Patients with progressive disease may cross over to arm II after at least 4 months on study and up to 1 year from the time of randomization. Patients who cross over receive erythropoietin alone.
* Arm II (Erythropoietin): Patients receive erythropoietin subcutaneously (SC) or intravenously (IV) daily. Patients undergo bone marrow aspirate and biopsy as in arm I. Treatment continues daily for a maximum of 1 year.

Patients with stable or progressive disease at day 120 receive filgrastim (G-CSF) SC daily or 3 days a week and erythropoietin SC daily for up to 6 months. Patients with no response to G-CSF and lower-dose erythropoietin may proceed to a higher dose of erythropoietin.

Quality of life is assessed at baseline, every 4 months during study, and at study completion.

Patients are followed every 4 months for 2 years, every 6 months for 3 years, and then annually for 5 years.

ACTUAL ACCRUAL: A total of 118 patients were accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Diagnosis of a myelodysplastic syndrome
* Refractory anemia (RA)
* RA with ringed sideroblasts
* RA with excess blasts (RAEB). RAEB patients must have a bone marrow blast count of less than 20% and less than 5% blast forms on peripheral blood
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 3
* Platelet count greater than 30,000/mm^3 (without platelet transfusions)
* Hematocrit less than 30% (pretransfusion)
* Bilirubin less than 3 mg/dL
* Blood urea nitrogen (BUN) less than 40 mg/dL or Creatinine less than 2.0 mg/dL
* Prior epoetin alfa allowed provided dosage was less than 30,000 units per week for less than 1 month duration
* At least 1 month since prior erythropoietin
* At least 2 months since prior recombinant growth factor
* At least 2 months since prior chemotherapy for other malignancy or autoimmune disease
* At least 2 weeks since prior androgen or steroids for treatment of myelodysplastic syndromes

Exclusion Criteria:

* RAEB in transformation
* Chronic myelomonocytic leukemia
* Splenomegaly greater than 6 cm below the left costal margin or greater than 3 times normal size
* Uncontrolled hypertension
* Sensitivity to E. coli-derived proteins
* Sensitivity to epoetin alfa or any of its components (e.g., human albumin)
* Documented iron deficiency. If marrow iron stain is not available, the transferrin saturation must be greater than 20% or ferritin greater than 100 ng/dL
* Active infection or bleeding
* Other uncontrolled malignancy
* Pregnant or nursing. Fertile patients must use effective contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 1998-03-04 (Actual); Primary Completion 2008-08 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth B. Miller, MD, Study Chair — Beth Israel Deaconess Medical Center
Locations (28):
- United States (28):
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tufts - New England Medical Center, Boston, Massachusetts
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - MetroHealth's Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - CCOP - Scott and White Hospital, Temple, Texas
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin

REFERENCES:
- [Background] Cherry AM, Brockman SR, Paternoster SF, Hicks GA, Neuberg D, Higgins RR, Bennett JM, Greenberg PL, Miller K, Tallman MS, Rowe J, Dewald GW. Comparison of interphase FISH and metaphase cytogenetics to study myelodysplastic syndrome: an Eastern Cooperative Oncology Group (ECOG) study. Leuk Res. 2003 Dec;27(12):1085-90. doi: 10.1016/s0145-2126(03)00104-8. PMID 12921944
- [Result] Greenberg PL, Sun Z, Miller KB, Bennett JM, Tallman MS, Dewald G, Paietta E, van der Jagt R, Houston J, Thomas ML, Cella D, Rowe JM. Treatment of myelodysplastic syndrome patients with erythropoietin with or without granulocyte colony-stimulating factor: results of a prospective randomized phase 3 trial by the Eastern Cooperative Oncology Group (E1996). Blood. 2009 Sep 17;114(12):2393-400. doi: 10.1182/blood-2009-03-211797. Epub 2009 Jun 29. PMID 19564636
- [Result] Miller KB, Kim HT, Greenberg P, et al.: Phase III prospective randomized trial of EPO with or without G-CSF versus supportive therapy alone in the treatment of myelodysplastic syndromes (MDS): results of the ECOG- CLSG trial (E1996). [Abstract] Blood 104 (11): A-70, 2004.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on December 9, 1997, accrued its first patient on March 4, 1998, and closed on June 1, 2004. A total of 118 patients were enrolled (110 ECOG patients and 8 Canadian Leukemia Study Group [CLSG] patients).
Period: Step 1
Arm/Group | Supportive Care | Erythropoietin
Started | 61 | 57
Patients With Complete Data | 57 | 53
Treated | 56 | 53
Eligible and Treated | 52 | 50
Patients With QOL Data at 4 Months | 42 | 42
Patients With Transfusion Data | 37 | 42
Completed | 0 | 0
Not Completed | 61 | 57
Not completed — Reasons off treatment not documented | 60 | 57
Not completed — Never started treatment | 1 | 0
Period: Step 2 (Cross Over)
Arm/Group | Supportive Care | Erythropoietin
Started | 26 | 0 (Only patients in the supportive care arm are eligible to cross over to the Erythropoietin arm.)
Completed | 0 | 0
Not Completed | 26 | 0
Not completed — Reasons off treatment not documented | 26 | 0
Period: Step 3 (EPO 150 Units/kg and G-CSF)
Arm/Group | Supportive Care | Erythropoietin
Started | 12 | 20
Treated | 12 | 19
Completed | 0 | 0
Not Completed | 12 | 20
Not completed — Off treatment reasons not documented | 12 | 19
Not completed — Never started treatment | 0 | 1
Period: Step 4 (EPO 300 Units/kg and G-CSF)
Arm/Group | Supportive Care | Erythropoietin
Started | 6 | 7
Completed | 0 | 0
Not Completed | 6 | 7
Not completed — Off treatment reasons not documented | 6 | 7

BASELINE CHARACTERISTICS:
Population: All patients with complete data are included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Supportive Care | Erythropoietin | Total
Number analyzed (Participants) | 57 | 53 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 10 | 17
  >=65 years | 50 | 43 | 93
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 41
  Male | 36 | 33 | 69

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Free of Transfusion at 4 Months
Description: Whether a patient required transfusion or not at 4 months was recorded.
Time Frame: Assessed at 4 months
Population: Only patients with transfusion data were included in this analysis.
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Arm/Group | Supportive Care | Erythropoietin
Number analyzed (Participants) | 37 | 42
Proportion of patients | 0.459 [0.295 to 0.631] | 0.714 [0.554 to 0.843]

2. Secondary Outcome: Overall Survival
Description: Time from randomization to death from any cause. Patients alive at the time of analysis were censored at the date of last contact.
Time Frame: Assessed every 3 months for 2 years, every 6 months for 3 subsequent years, and annually thereafter
Population: All patients with complete data were included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Supportive Care | Erythropoietin
Number analyzed (Participants) | 57 | 53
Months | 31 [23.5 to 48.0] | 37 [24.4 to 40.8]

3. Secondary Outcome: Quality of Life- Total Functional Assessment of Cancer Therapy - General (FACT-G) Score at 4 Months
Description: The FACT-G scale has 4 dimensions, including physical well-being, social/family well-being, emotional well-being, and functional well-being. The score for each subscale was added together to obtain the total FACT-G score that was evaluated on this study. The total FACT-G score ranges from 0 to 108 with higher scores reflecting better quality of life. It was administered at the time of study entry, every 4 months for the first year, and at the time patient went off treatment. Due to limited data after 4 months on treatment, the analysis was restricted to the four-month time point.
Time Frame: Assessed at 4 months
Population: Only patients who completed quality of life assessment at 4 months were included in this analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Supportive Care | Erythropoietin
Number analyzed (Participants) | 42 | 42
Scores on a scale | 84.1 (15.77) | 84.33 (14.75)

ADVERSE EVENTS:
Time Frame: Adverse events were reported within 10 days of any reportable events specified in the protocol while on treatment and for 30 days after the end of treatment.
Groups:
- Supportive Care (Step 1): Patients received red cell and platelet transfusions for symptoms or to maintain hematocrit at or above 25% by volume. Patients who required transfusion support for symptomatic anemia prior to entering the study and who developed an increase in their transfusion requirement of >= 50% shall cross over to the Erythropoietin treatment arm, after at least four months on the supportive therapy arm.
- Erythropoietin (Step 1): Erythropoietin was administered at 150 units/kg subcutaneously every day. If patients stopped responding, they were subsequently treated with Erythropoietin (150 units/kg) and filgrastim and then Erythropoietin (300 units/kg) and filgrastim.
- Erythropoietin (Cross-over; Step 2): Patients in the supportive care arm who required transfusion support for symptomatic anemia prior to entering the study and who developed an increase in their transfusion requirement of >= 50% shall cross over to the Erythropoietin treatment arm, after at least four months on the supportive therapy arm. Erythropoietin was administered at 150 units/kg subcutaneously every day.
- Erythropoietin (150 Units/kg) and Filgrastim (Step 3): All patients received erythropoietin alone treatment may, at progression or at stable disease with continued transfusion requirement following 4 months of therapy, add filgrastim.
- Erythropoietin (300 Units/kg) and Filgrastim (Step 4): All patients received erythropoietin (150 units/kg) and filgrastim may, at progression or at stable disease with continued transfusion requirement following 4 months of therapy, increased their dose of erythropoietin to 300 units/kg.
Arm/Group | Supportive Care (Step 1) | Erythropoietin (Step 1) | Erythropoietin (Cross-over; Step 2) | Erythropoietin (150 Units/kg) and Filgrastim (Step 3) | Erythropoietin (300 Units/kg) and Filgrastim (Step 4)
Serious Adverse Events (participants affected / at risk) | 0/56 | 16/53 | 7/26 | 6/31 | 1/13
Other Adverse Events (participants affected / at risk) | 8/56 | 28/53 | 13/26 | 18/31 | 8/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Supportive Care (Step 1) (N=56) | Erythropoietin (Step 1) (N=53) | Erythropoietin (Cross-over; Step 2) (N=26) | Erythropoietin (150 Units/kg) and Filgrastim (Step 3) (N=31) | Erythropoietin (300 Units/kg) and Filgrastim (Step 4) (N=13)
Anemia (Blood and lymphatic system disorders) | 0 | 3 | 2 | 3 | 0
Hemorrhage (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 2 | 3 | 1 | 0
Fever w/o infection (General disorders) | 0 | 1 | 0 | 0 | 0
GU adverse event (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Liver (Gastrointestinal disorders) | 0 | 8 | 2 | 1 | 0
Cardiac adverse event (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Neuropathy-sensory (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Metabolic (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 1 | 1 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Impotence (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Other toxicities (General disorders) | 0 | 1 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Supportive Care (Step 1) (N=56) | Erythropoietin (Step 1) (N=53) | Erythropoietin (Cross-over; Step 2) (N=26) | Erythropoietin (150 Units/kg) and Filgrastim (Step 3) (N=31) | Erythropoietin (300 Units/kg) and Filgrastim (Step 4) (N=13)
Hemorrhage (Blood and lymphatic system disorders) | 0 | 3 | 2 | 2 | 1
Infection (Infections and infestations) | 0 | 8 | 0 | 1 | 2
GU adverse event (Renal and urinary disorders) | 0 | 6 | 1 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 9 | 5 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 4 | 2 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 10 | 3 | 2 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 3 | 1 | 0 | 0
Liver (Gastrointestinal disorders) | 0 | 5 | 0 | 6 | 0
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 2 | 3 | 3
Skin (Skin and subcutaneous tissue disorders) | 0 | 10 | 3 | 1 | 1
Weight loss (Investigations) | 1 | 3 | 3 | 2 | 1
Neuropathy-sensory (Nervous system disorders) | 0 | 3 | 0 | 0 | 0
Neuropathy-clinical (Nervous system disorders) | 1 | 11 | 1 | 2 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 6 | 3 | 1 | 0
Epigastric distress (Gastrointestinal disorders) | 0 | 5 | 0 | 1 | 0
Edema (General disorders) | 0 | 6 | 2 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 1 | 0
Fatigue (General disorders) | 4 | 12 | 8 | 10 | 4
Cardiac adverse event (Cardiac disorders) | 0 | 1 | 4 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 2 | 1
Fever w/o infection (General disorders) | 0 | 1 | 1 | 2 | 0
Neuropathy-psych (Nervous system disorders) | 0 | 1 | 1 | 2 | 1
Abdominal cramps (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Hot flashes (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No